CLINICAL TRIAL: NCT00900081
Title: Evaluation of Cyclooxygenase-2 Expression in Normal Cervix, Cervical Intraepithelial Neoplasia and Early Invasive Squamous Cell Carcinoma With Correlation to Parameters of Invasion and Angiogenesis
Brief Title: Cyclooxygenase-2 Expression in Tissue Samples From Patients With a Normal Cervix, Cervical Intraepithelial Neoplasia, or Early Invasive Cervical Cancer
Status: Withdrawn | Type: Observational
Why Stopped: no accrual, PI left institution
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000550067; CCCWFU-00A03; CCCWFU-BG01-137
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2015-10

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical squamous cell carcinoma; stage IA cervical cancer; stage 0 cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of tissue from patients with or without cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This laboratory study is looking at cyclooxygenase-2 expression in tissue samples from patients with a normal cervix, cervical intraepithelial neoplasia, or early invasive cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine cyclooxygenase-2 (COX-2) levels in biopsy or surgical specimens from patients with normal cervical epithelium, cervical intraepithelial neoplasia, or microinvasive squamous cell carcinoma of the cervix.
* Correlate COX-2 levels with histological diagnosis and parameters of invasion (i.e., matrix metalloproteinase, microvessel count, and VEGF).

OUTLINE: Paraffin-embedded tissue samples are analyzed by immunohistochemistry for evaluation of cyclooxygenase-2 levels, microvessel count, and matrix metalloproteinase and VEGF expression.

Medical data for study analysis is obtained by retrospective review of patient charts.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Underwent hysterectomy with removal of a normal cervix for diagnosis unrelated to cancer or cervical dysplasia
  * Underwent cervical biopsy or removal of cervical tissue and diagnosed with cervical intraepithelial neoplasia (CIN) grades 1-3
  * Underwent cervical biopsy and diagnosed with microinvasive squamous cell carcinoma of the cervix
* Paraffin-embedded tissue samples of normal cervical epithelium, CIN, or microinvasive squamous cell carcinoma of the cervix must be available for examination

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Cervical Intraepithelial Neoplasia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Cyclooxygenase-2 (COX-2) levels in cervical intraepithelial neoplasia (CIN) | day 1
Correlation of COX-2 levels in CIN with histological diagnosis and parameters of invasion | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte E. Miller, MD, Study Chair — Wake Forest University Health Sciences